CLINICAL TRIAL: NCT02301273
Title: Being Awake, Upright and Moving as the Basis for Early ICU Physiotherapy: Comparison of Patient Outcomes Between Enhanced and Conventional ICU Physiotherapy
Brief Title: Being Awake, Upright and Moving as the Basis for Early ICU Physiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Landspitali University Hospital (Other)
Collaborators: University of Iceland (Other)
Responsible Party: Principal Investigator, Olof Ragna Amundadottir, Principal Investigator, Landspitali University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16.2011
Record Dates: First submitted 2012-03-12; First posted 2014-11-25 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Critical Illness
Keywords: Intensive care unit; Physiotherapy; Upright position; Exercise; Long term follow up of ICU survivors
MeSH Terms: conditions — Critical Illness; Motor Activity | interventions — Intensive Care Units; Physical Therapy Modalities; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Physiotherapy (Active Comparator): Patients will receive the usual physiotherapy treatment in ICU in Iceland from day 5 after intubation, which adheres to international standards of practice, including the potential for no treatment. Usual physiotherapy once daily for 20 minutes.
  Interventions: Other: Usual Physiotherapy
- Enhanced Physiotherapy (Experimental): Patients will receive the intervention physiotherapy treatment consisting of exercises and a progressive upright positioning and mobilization (20 minutes) twice daily from day 3 (>48 hours) after intubation including the potential for no treatment, if they are stable, even though they are not completely alert, Total treatment time of 40 minutes.
  Interventions: Other: Enhanced Physiotherapy

INTERVENTIONS:
Other: Usual Physiotherapy — o Patients will receive the usual physiotherapy treatment in ICU in Iceland from day 5 after intubation, which adheres to international standards of practice, including the potential for no treatment. Usual physiotherapy once daily for 20 minutes.
  Other Names: Intensive care unit; Physiotherapy; Long term follow up of ICU survivors
  Arms: Usual Physiotherapy
Other: Enhanced Physiotherapy — o Patients will receive the intervention physiotherapy treatment consisting of exercises and a progressive upright positioning and mobilization (20 minutes) twice daily from day 3 (>48 hours) after intubation including the potential for no treatment, if they are stable, even though they are not completely alert, Total treatment time of 40 minutes.
  Other Names: Intensive care unit; Physiotherapy; Upright position; Exercise; Long term follow up of ICU survivors
  Arms: Enhanced Physiotherapy

SUMMARY:
Patients who have been admitted to Intensive Care Units (ICU) and are intubated and mechanically ventilated for longer than 48 hours have impaired physical, psychological and social health and well-being six to twelve months after discharge. The advocacy of intensive physiotherapy and mobilization early in the course of critical illness has been established. It is of great importance to study the long-term outcomes (physical function and quality of life) in intubated and ventilated patients who start exercising and ambulating mobilizing) as soon as possible during ICU stay because the most effective mode, intensity or frequency of exercise needs to be identified.

The aim is to study the short- and long-term outcomes of enhanced early physiotherapy and upright position in critically ill patients on prolonged invasive ventilation and to develop principles to guide physiotherapists in their clinical decision making in the ICU.

DETAILED DESCRIPTION:
Mobilization is an intervention prescribed by physiotherapists, for critically ill patients in the ICU, to prevent as well as remediate a range of multisystem problems and complications. Mobilization which refers to low levels of exercise and progressive position changes from being supine to being upright and moving, is both a gravitational and an exercise stimulus. Given the hemodynamic status of patients in the ICU can change suddenly, physiotherapists gauge the patient's status moment by moment, and change the parameters of an intervention accordingly, i.e., the type and level of an intervention, its duration and rest periods. The aim of this research is to study the short- and long-term outcomes of enhanced early physiotherapy, with mobilization and upright position, in critically ill patients on prolonged invasive ventilation. This is a prospective, randomized, single blind trial where the intervention permits variation in the physiotherapist's clinical decision making to simulate the general practice. This study started in November 2011, data collection and intervention will continue until November 2014 with 12 months follow up until november 2015.

ELIGIBILITY:
Inclusion Criteria:

* Patient participants will be at least 18 years of age and admitted to the ICU of Landspitali Fossvogur or Landspitali Hringbraut of the The National University Hospital of Iceland.
* Intubated and on mechanical ventilation for > 48 hours
* Icelandic speaking.
* Upright position and ambulation is not contraindicated or impossible.

Exclusion Criteria:

-Those patients deemed by the medical teams of each unit not to be sufficiently stable. These would include diagnoses such as: Intracranial insults including:Severe head injury, Subarachnoidal hemorrhage, Elevated intracranial pressure, Intraventricular drain, Neurological deterioration, Status epileptics

* Unstable fractures of the vertebral column
* Spinal cord injuries
* Unstable pelvic fractures and/or balanced skeletal traction
* Severe burns
* Mental status precluding being able to follow instructions and cooperate with treatment appropriately

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Length of ICU and hospital stay | ICU discharge an expected average of 7 days / hospital discharge an expected average of 21 days
  Length of ICU and hospital stay will be measured in days and hours

SECONDARY OUTCOMES:
Physical Function | ICU discharge an expected average of 7 days / hospital discharge an expected average of 21 days and 3, 6 and 12 months after ICU discharge
  Medical Research Council - sum-score
Physical function | ICU discharge an expected average of 7 days / hospital discharge an expected average of 21 days and 3, 6 and 12 months after ICU discharge
  Modified Barthel Index
Physical function | 3,6,12 months after discharge from ICU
  6 min walk test,
Health Related Quality of Life | 0,3,6,12 months after discharge from ICU
  Short Form-36v2,

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Dean, PhD, Study Chair — University of Iceland; Gísli H Sigurðsson, PhD, Study Chair — Landspítali University Hospital and University of Iceland; Þórarinn Sveinsson, PhD, Study Chair — University of Iceland; Helga Jónsdóttir, PhD, Study Chair — University of Iceland; Alma Möller, PhD, Study Chair — Landspítali University Hospital
Locations (1):
- Landspítali University Hospital, Reykjavik, Iceland